CLINICAL TRIAL: NCT02637479
Title: Treatment of Opioid-refractory Pain (WHO Level III) by Pituitary Radiosurgery: A Multicenter, Prospective, Randomized Study
Brief Title: Treatment of Opioid-refractory Pain (WHO Level III) by Pituitary Radiosurgery
Acronym: Hyporadoul
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-51; 2015-A00616-43 (Registry Identifier: IDRCB); RCAPHM15_0022 (Other: APHM)
Record Dates: First submitted 2015-12-15; First posted 2015-12-22 (Estimated); Last update posted 2025-01-30 (Actual); Status verified 2015-12

CONDITIONS: Any Cancer With Multiple Bone Metastases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pituitary radiosurgery group (Experimental): Subjects will receive a pituitary radiosurgery by GammaKnife® during a brief hospitalization associated with standards of care for pain according to recommendations (Standards, Options and Recommendations about drug analgesic treatments for nociceptive cancer pain in adults)
  Interventions: Device: GammaKnife®; Device: 18F-2-fluoro-2-deoxy-D-glucose - positron emission tomography (FDG-PET); Device: MRI
- Control group (Active Comparator): Subject will receive standards of care for pain according to recommendations (Standards, Options and Recommendations about drug analgesic treatments for nociceptive cancer pain in adults)
  Interventions: Device: 18F-2-fluoro-2-deoxy-D-glucose - positron emission tomography (FDG-PET)

INTERVENTIONS:
Device: GammaKnife®
  Arms: Pituitary radiosurgery group
Device: 18F-2-fluoro-2-deoxy-D-glucose - positron emission tomography (FDG-PET)
Device: MRI
  Arms: Pituitary radiosurgery group

SUMMARY:
80% of palliative care cancer patients suffer from severe pain. The management of these pain improves the quality of life of these patients. The management of opioid pain refractory to date remains a difficulty for caregivers. Hypophysectomy performed to try to control hormone-dependent neoplasia also help relieve pain associated with lesions secondary cancer. The surgical hypophysialis radio Gamma Knife ® was recently performed on a small number of patients. She would have the advantage of reducing the risk of complications compared to other techniques and achieve similar analgesic effect on diffuse, or mixed nociceptive pain associated with metastases on average in 2 days and would reduce or stop opiates most often responsible for side effects impairing the quality of life. The objective of this clinical trial, multicenter, prospective, randomized controlled is to evaluate the effectiveness of surgical hypophysialis radio for patients in palliative situations with refractory cancer pain in opioid level III. The type of pain "cancer pain" was done in order to optimize the recruitment and homogenization of the study population: patients cared for in palliative care units are mostly patients cancer (70-80%). This study is therefore part of a palliative setting and the results of this test can be extrapolated to other populations of palliative patients with refractory pain.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman, aged 18 years or older;
* Subject suffering from nociceptive or mixed pain, not related to acts, refractory to standard opioid therapy
* Subject having a cancer defined by histology whatever the origin of the primitive cancer,
* Subject having multiple bone metastases
* Subject in palliative care state according to the definition given by the French Society of Palliative Care and Support
* Subject supported by structures of palliative care, pain or cancer involved in the study
* Inpatient and outpatient
* Subject without a curative cancer treatment and with or without palliative anticancer treatment;
* Subject non in "ultimate" phase (estimated survival superior at 48 h by a physician)
* Subject with acceptable general condition (Karnofsky performance Status Scale superior at 40
* Subject with a preserved vigilance defined from the Epworth scale
* Subject with preserved cognition according to the scale Basic Test Concentration, Memory and Guidance (TELECOM)
* Subject which can fill in a questionnaire, able to read or to understand the French language;
* Subject who signed an informed consent;
* Subject affiliated to the French health insurance system.

Exclusion Criteria:

* Subject with a curative cancer treatment
* Subject in "ultimate" phase (estimated by the physician of survival less than 48 hours)
* History of whole brain radiation
* History of radiosurgery of pituitary lodge
* Subject treated there less than a month by external or metabolic radiotherapy analgesic, surgical analgesic technic
* Subject minor, pregnant or breastfeeding, subject not being affiliated to the French health insurance system or private about freedom;
* Subject refusing to participate in the study or not signing the informed consent.
* Subject allergic to any component of Fludeoxyglucose (18F)
* Subject allergic to gadolinium salts.
* Subject with severe renal impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-12; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The pain assessment | 36 months
  using the Numeric Pain Intensity Scale (NPSI)
The pain assessment | 36 months
  Neuropathic pain questionnaire (DN4)
The pain assessment | 36 months
  Self-reported pain and Quality of life

SECONDARY OUTCOMES:
assessment of the visual fields | 36 months
  visual perimeter test
assessment of the visual acuity | 36 months
  exploration test macular function
endocrine balance | 36 months
  Rate of Corticotropic in the blood
endocrine balance | 36 months
  Rate of Gonadotropic in the blood
endocrine balance | 36 months
  Rate of Somatotropic in the blood
endocrine balance | 36 months
  Rate of Thyrotropic in the blood
Pituitary morphology | 36 months
  MRI with gadolinium
evaluate metabolic consumption of glucose | 36 mois
  FDG-PET
evaluate metabolic connectivity at resting-state | 36 mois
  18F-2-fluoro-2-deoxy-D-glucose - positron emission tomography (FDG-PET)

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France